CLINICAL TRIAL: NCT00185601
Title: Internet Diabetes Self-Management Evaluation
Brief Title: Internet Diabetes Self-Management Workshop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kate Lorig, professor emertius, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 5R18DK065729-02 (NIH)
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- on-line self management intervention (Other)
  Interventions: Behavioral: Internet Diabetes Self-Management Program
- usual care control group (No Intervention)
- on-line self management intervention with email reinforcement (Experimental)
  Interventions: Behavioral: Internet Diabetes Self-Management Program

INTERVENTIONS:
Behavioral: Internet Diabetes Self-Management Program
  Arms: on-line self management intervention; on-line self management intervention with email reinforcement

SUMMARY:
The purpose of this study is to determine of the effectiveness of an Internet based Diabetes Self-Management workshop for people with type II diabetes. Half of the people who complete the workshop will be invited to continue their education by participating in a email discussion group. Thus, we will be able to learn both the efficacy of the original program as well as its efficacy when reinforced by the discussion group.

Diabetes is a disease that must be managed day by day by the individual with the disease. Although we know a great deal about the self-management of type II diabetes, most self-management is less than optimal. In addition, most people with diabetes do not have an opportunity to participate in formal diabetes education. This study will determine if an Internet delivered educational workshop will help people with diabetes manage their disease. Thus we will be measuring changes in behaviors, changes in symptoms and changes in HbA1c, blood pressure, cholesterol, and weight. If successful the workshop will serve as a prototype for Internet diabetes education.

ELIGIBILITY:
Inclusion Criteria::- Diabetes type 2

* Have internet access and email address
* Live in the United States
* 18 years of age or older Exclusion Criteria:- Previous participation in similar online or community-based self-management program
* Active treatment for cancer
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 761 (Actual)
Dates: Start 2006-02; Primary Completion 2009-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
HbA1c | 6 and 12 months

SECONDARY OUTCOMES:
Outcome Measure: Health-related quality of life | 6 and 12 months
Outcome Measure: Health behaviors | 6 and 12 months
Health care utilization | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kate R Lorig, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Case S, Jernigan V, Gardner A, Ritter P, Heaney CA, Lorig KR. Content and frequency of writing on diabetes bulletin boards: does race make a difference? J Med Internet Res. 2009 Jun 24;11(2):e22. doi: 10.2196/jmir.1153. PMID 19632975